CLINICAL TRIAL: NCT02638324
Title: Supportive Treatment of Severe Heart Failure by Renal Denervation
Acronym: Heart-RND
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of the lack of the candidates and because of restrictions of denervation at the completion date.
Sponsor: Turku University Hospital (Other Government)
Collaborators: Satakunta Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Juhani02
Record Dates: First submitted 2015-05-20; First posted 2015-12-23 (Estimated); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Heart Failure
Keywords: Renal nervous denervation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Renal nervous denervation. (Active Comparator): Renal nervous denervation is performed to the patients who do not response properly to conventional therapy. The patients are randomised according to the waiting list principle.
  Interventions: Procedure: Renal nervous denervation
- Renal nervous denervation (delayed) (Active Comparator): Renal nervous denervation is performed after six months on the waiting list
  Interventions: Procedure: Renal nervous denervation

INTERVENTIONS:
Procedure: Renal nervous denervation — The heart failure patients will undergo renal nervous denervation if they have not properly responded to medication and biventricular pacing therapy.

SUMMARY:
The overactivity of sympathetic nervous system is worsening the hemodynamic state of heart failure patients. The present study is planned to reduce the sympathetic tone in patients with severe heart failure by renal nervous denervation.

DETAILED DESCRIPTION:
The patient population consists of heart failure patients who are not responding properly to medication and biventricular pacing therapy. The inappropriate response to these therapies is evaluated by patient history (NYHA III-IV), echocardiography (EF < 45%), 6-minute walking test (<440m) and measurements of P-ProBNP. The patients who fulfill the inclusion criteria will undergo renal nervous denervation. The patients will be followed up with the same methods as they were recruited to the study (by patient history (NYHA III-IV), echocardiography (EF < 45%), 6-minute walking test (<440m) and measurements of P-ProBNP). The overall time of follow-up will be 24 months. The patients are randomised according to the waiting list principle in a manner to 1:1. The waiting time will be 6 months.

ELIGIBILITY:
Inclusion Criteria:

* NYHA III-IV
* ejection fraction <45 %
* 6-minute walking test under 440m

Exclusion Criteria:

* Unstable hemodynamic state
* uncooperation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
6-minute walking test | 24 months
  Composite outcome measure

SECONDARY OUTCOMES:
Patient history | 24 months
  Composite outcome measure
Cardiac echocardiography | 24 months
  Composite outcome measure
P-proBNP | 24 months
  Composite outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Mari-Anne Vaittinen, MD, Study Chair — Vaasa Central Hospitla; Mari-Anne Vaittinen, MD, Study Chair — Vaasa Central Hospital, Vaasa, Finland
Locations (1):
- Vaasa Central Hospital, Vaasa, Finland